CLINICAL TRIAL: NCT03415516
Title: Clinical Comparison of Universal Adhesives in Terms of Different Application Modes on the Restoration of NCCLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universal Clinical NCCLs
Record Dates: First submitted 2017-12-23; First posted 2018-01-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Tooth Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Gluma Universal, self-etch mode (GSE) (Experimental)
  Interventions: Device: Gluma Universal
- Gluma Universal, selective etching (GSL) (Experimental)
  Interventions: Device: Gluma Universal
- Gluma Universal, etch&rinse (GER) (Experimental)
  Interventions: Device: Gluma Universal
- All Bond Universal, self-etch (ASE) (Experimental)
  Interventions: Device: All Bond Universal
- All Bond Universal, selective etching (ASL) (Experimental)
  Interventions: Device: All Bond Universal
- All Bond Universal, etch&rinse (AER) (Experimental)
  Interventions: Device: All Bond Universal
- Single Bond2, etch&rinse (SBU) (Experimental)
  Interventions: Drug: Single Bond2

INTERVENTIONS:
Device: Gluma Universal — Adhesive systems
  Arms: Gluma Universal, etch&rinse (GER); Gluma Universal, selective etching (GSL); Gluma Universal, self-etch mode (GSE)
Device: All Bond Universal — Adhesive systems
  Arms: All Bond Universal, etch&rinse (AER); All Bond Universal, selective etching (ASL); All Bond Universal, self-etch (ASE)
Drug: Single Bond2 — Adhesive systems
  Arms: Single Bond2, etch&rinse (SBU)

SUMMARY:
The aim of this randomized, controlled, prospective clinical trial is to evaluate the performances of two different universal adhesives and an etch&rinse adhesive in restoration of non-caries cervical lesions. Twenty patients will receive restorations. Lesions will be divided into 7 groups according to adhesive systems and application modes: GSE: Gluma Universal- self etch, GSL: Gluma Universal-selective etching, GER: Gluma Universal-etch&rinse, ASE: All Bond Universal- self etch, ASL: All Bond Universal- selective etching, AER: All Bond Universal- etch&rinse, SB (Control): Single Bond2+etch&rinse. Restorations (nano-hybrid composite) will be scored with regard to retention, marginal discoloration, marginal adaptation, recurrent caries and post operative sensitivity using modified USPHS criteria after 48 months. Two examiners who is not involved in the placement of restorations will conduct the evaluations. Descriptive statistics will be performed using Chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be as follows:

1. being 18 years or older,
2. having no medical or behavioral problems preventing then from attending review visits,
3. having at least 7 tooth with NCCLs (d) having antagonist teeth.

Exclusion Criteria:

Exlusion criteria will be:

1. poor gingival health,
2. uncontrolled, rampant caries,
3. bruxism,
4. removable partial dentures,
5. xerostomia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical performances of different adhesives | Two years
  Two year examinations according to USPHS criteria